CLINICAL TRIAL: NCT02064608
Title: A Phase 1 Window of Opportunity Study Investigating the Pharmacodynamic Biomarker Effects of AZD2014 (an mTOR1/2 Inhibitor) Given Prior to Radical Prostatectomy
Brief Title: Investigating the Effects of AZD2014 Therapy Given Prior to Radical Prostatectomy in Men With High Risk Prostate Cancer
Acronym: CaNCaP02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, CCTU- Cancer Theme, Cambridge Clinical Trials Unit - Cancer Theme, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CANCAP02; 2014-000214-56 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Prostate Cancer; High Risk; Intermediate Risk; Early disease; Neoadjuvant treatment; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Disease | interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD2014 (Experimental): This is a single arm study whereby a cohort of 20 patients with early high risk prostate cancer will be treated with a 15-day course of AZD2014 (mTOR inhibitor) treatment prior to radical prostatectomy.
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014 — mTOR inhibitor
  Other Names: AZ12729279

SUMMARY:
Patients with localised prostate cancer can be treated by radical prostatectomy (prostate gland removal surgery) or radiotherapy. Around 15% of men with prostate cancer are diagnosed with high risk disease meaning they are more likely to suffer treatment failure, disease progression and mortality. To date little progress has been made towards identifying effective treatment strategies that might delay or prevent disease recurrence in this patient population. Better identification of patients at high risk of relapse and improvements in therapy are therefore research priorities.

A protein named Mammalian Target of Rapamycin (mTOR) is known to play an important role in the development of prostate cancer. mTOR forms two protein complexes (mTORC1 and mTORC2) and sends signals helping cancer cells to grow while controlling their energy use. Blocking the function of mTOR, with an inhibitor such as AZD2014, might shut down the supply of energy supply to tumour cells leading to reduced cell growth and potentially slowing the progression of the disease.

The purpose of this study is to investigate the molecular pharmacology of AZD2014 treatment given to patients with prostate cancer prior to radical prostatectomy. The feasibility, safety and tolerability of a short course of AZD2014 will also be assessed.

DETAILED DESCRIPTION:
Eligible patients will be required to take 50mg AZD2014 tablets twice daily for 15 days prior to radical prostatectomy.

Immunohistochemistry will be carried out on prostate tumour biopsies taken at baseline and at radical prostatectomy in order to detect phosphorylated biomarkers of mTOR signalling and determine the amount of mTORC1 and mTORC2 signalling inhibition caused by AZD2014 treatment.

On the day of radical prostatectomy, blood samples will be collected pre- and at specified times post- dose for pharmacokinetic analyses.

Additional blood samples will be collected to study any genetic changes to the DNA, RNA and circulating tumour DNA (ctDNA) which may have been caused by AZD2014 treatment.

Refer to the "outcome measures" section for further information.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years old or older
* ECOG performance status of 0 or 1
* Clinical diagnosis of Intermediate (one or more of stage T2, or PSA >10ng/mL, or Gleason score of at least 7) or High Risk Prostate Cancer (one or more of stage T2c, or PSA >20ng/mL, or Gleason score of at least 8)
* Patient suitable for radical prostatectomy, following discussion at specialist MDT and subsequent review by surgical team
* Willing to use barrier contraceptive method, e.g. condom & spermicide
* Adequate bone marrow reserve or organ function (as specified in the study protocol)
* Normal chest radiograph and oxygen saturations, OR normal CT thorax

Exclusion Criteria:

* Contraindication to AZD2014 (as specified in the study protocol)
* Patients who have experienced any of the following procedures in the past 12 months: coronary artery bypass graft; angioplasty; vascular stent; myocardial infarction; angina pectoris; congestive heart failure (New York Heart Association grade of 2 or above); ventricular arrhythmias requiring continuous therapy; supraventricular arrhythmias including atrial fibrillation, which are uncontrolled; haemorrhagic or thrombotic stroke including transient ischaemic attacks or any other CNS bleeding.
* Previous chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents and/or investigational agents within 28 days of starting study treatment.
* Major surgery within 4 weeks prior to study entry (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study
* Potent or moderate inhibitors and inducers of CYP2C8 if taken within the stated wash-out period: Gemfibrozil, trimethoprim, glitazones, montelukast, deferasirox and quercetin (1-week minimum wash out period)
* Any haematopoietic growth factors, e.g. G-CSF, GM-CSF, within 4 weeks prior to receiving study drug
* As judged by the Investigator, any evidence of severe or uncontrolled systemic disease (as specified in the study protocol)
* Abnormal ECHO or MUGA at baseline
* Mean resting QTc of 470msec or above (as per local reading)
* Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation, or risk of arrythmic events (examples specified in study protocol). History of Torsades de Pointes.
* Patients with Diabetes Type I or uncontrolled Type II as judged by the investigator
* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
* Unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
To measure the amount of inhibition (percentage change from baseline) in mTORC1 and mTORC2 signalling in tumour samples from men with early, high-risk prostate cancer after AZD2014 treatment | 2 weeks
  Participants will be treated with AZD2014 for 15 days prior to radical prostatectomy surgery. To assess the amount of mTORC1 and mTORC2 inhibition caused by AZD2014 treatment, phosphorylated signalling biomarkers (namely p4EBP1, pS6 and pAKT) will be detected by immunohistochemistry and quantified. The amount of mTORC1 and mTORC2 signalling inhibition will be determined by comparison of prostate tumour biopsies taken at baseline (time of diagnosis) and following AZD2014 treatment. An intra-operative prostate biopsy will also be taken in order to evaluate variability between samples.

SECONDARY OUTCOMES:
To determine the incidence of adverse events due to AZD2014 given prior to radical prostatectomy | 8 weeks unless further observation is clinically indicated
  In order to assess the safety and feasibility of AZD2014 treatment prior to radical prostatectomy, a record will be kept of all adverse events experienced by the participants. Adverse events will be detailed by the study team when the participant attends inpatient/outpatient hospital visits and the participant will also be required to document their adverse events in a patient diary. Adverse events will be recorded for the duration of study treatment and for six weeks following treatment.
To determine the severity of adverse events due to AZD2014 prior to radical prostatectomy | 8 weeks unless further observation is clinically indicated
  The severity of all adverse events will graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

OTHER OUTCOMES:
To determine blood plasma concentration and pharmacokinetics of AZD2014. | Following 15 days AZD2014 treatment
  On the day of radical prostatectomy surgery, participants will have up to four blood samples taken before and after their AZD2014 dose for pharmacokinetic analysis. These samples will be used to construct a concentration-time curve for AZD2014 in the blood.
To measure the biological effects of AZD2014 treatment | Following 15 days AZD2014 treatment
  Participants will be treated with AZD2014 for 15 days prior to radical prostatectomy surgery. The biological effects of AZD2014 treatment will be determined by analysis of prostate tumour biopsies and blood samples taken at baseline and following AZD2014 treatment.
Exploratory endpoints | Following 15 days AZD2014 treatment
  The biological effects of AZD2014 on blood and prostate tumour samples will be investigated:
  Histological markers of tumour cell proliferation, apoptosis and androgen receptor control of tumour metabolism will be measured.
  Blood samples will be used to identify genetic changes in DNA, RNA and circulating tumor DNA caused by AZD2014 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Simon C Pacey, MRCP, PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No